CLINICAL TRIAL: NCT01326104
Title: Recurrent Medulloblastoma and Primitive Neuroectodermal Tumor Adoptive T Cell Therapy During Recover From Myeloablative Chemotherapy and Hematopoietic Stem Cell Transplantation
Brief Title: Vaccine Immunotherapy for Recurrent Medulloblastoma and Primitive Neuroectodermal Tumor
Acronym: Re-MATCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201500502; W81XWH-10-1-0089 (Other Grant/Funding Number: Department of Defense); CDMRP-PRO93877 (Other: Department of Defense); OCR13166 (Other: University of Florida)
Record Dates: First submitted 2010-07-22; First posted 2011-03-30 (Estimated); Results first posted 2022-02-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Medulloblastoma; Neuroectodermal Tumor
Keywords: Medulloblastoma; Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Medulloblastoma; Neuroectodermal Tumors; Neuroectodermal Tumors, Primitive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): High dose chemotherapy plus peripheral blood stem cell transplant followed by TTRNA-xALT and TTRNA-DCs.
  Interventions: Biological: TTRNA-xALT; Biological: TTRNA-DCs
- Group B (Experimental): NMA Salvage chemotherapy plus peripheral blood stem cell transplant followed by TTRNA-xALT and TTRNA-DCs.
  Interventions: Biological: TTRNA-xALT; Biological: TTRNA-DCs

INTERVENTIONS:
Biological: TTRNA-xALT — TTRNA-xALT 3 x 10^7/kg by intravenous injection once.
Biological: TTRNA-DCs — TTRNA-DCs 1 x 10^7 by intradermal injection every 2 weeks for 3 total doses.

SUMMARY:
Immunotherapy is a specific approach to treating cancer that has shown promise in adult patients for the treatment of melanoma, malignant brain tumors, and other cancers. The study investigators will use the experience they have gained from these studies to try to improve the outcome for children affected by a recurrent brain tumor.

Approximately 35 patients with first recurrence of medulloblastoma (reMB)/supratentorial primitive neuroectodermal tumors (PNETs) will be treated with tumor-specific immune cells and dendritic cell vaccines to see what impact they have on the tumor.

DETAILED DESCRIPTION:
Malignant brain tumors now represent the most frequent cause of cancer death in children. Despite aggressive and highly toxic multi-modality therapy including surgery, craniospinal radiation, and high-dose chemotherapy coupled with peripheral blood stem cell transplantation, almost half the children diagnosed with the most common malignant brain tumors, medulloblastoma (MB) and primitive neuroectodermal tumors (PNET), will still die from recurrent disease. Furthermore, survivors are often left with severe and lifelong treatment-associated cognitive and motor deficits. The development of more effective and tumor-specific therapies that will not add further toxicity to existing treatments is paramount in improving clinical outcomes for children affected by MB/PNETs. Immunotherapy targeting tumor-specific antigens expressed within brain tumors is a modality potentially capable of meeting this clear and urgent need.

Despite considerable advancements and promising clinical results observed in immunotherapy trials directed against adult malignant brain tumors, efforts in the immunologic treatment of pediatric brain tumors have been limited to relatively few notable studies. This is due, at least in part, to the often limited viable tumor tissue available for tumor cell-based vaccine preparations, and the lack of identification of consistently expressed tumor-specific antigens within these cancers.

The use of total tumor RNA (TTRNA)-loaded dendritic cells (DCs) was pioneered at Duke University, as a novel platform for inducing potent immunologic responses against the variety of uncharacterized and patient-specific antigens present within malignant tumor cells. Duke demonstrated that sufficient RNA for clinical vaccine preparations can be amplified with high fidelity using existing molecular technologies from as few as 500 isolated pediatric and adult brain tumor cells, thus allowing vaccine preparation from surgical biopsies and even microdissected archival tumor specimens.

Immunotherapy administered during recovery from chemotherapy may have tremendous advantages, as adoptive cellular therapy following lymphodepletive conditioning regimens has emerged as the most effective treatment strategy for advanced and refractory melanoma. Our hypothesis is that DC + ex vivo expanded Autologous Lymphocyte Transfer (xALT) therapy targeting recurrent MB/PNETs during recovery from myeloablative chemotherapy will be safe and will prolong survival in children and young adults with recurrent MB/PNETs.

In this study, the investigators will treat patients with first recurrence reMB/PNETs after completion of definitive radiation therapy with autologous tumor-specific T cell immunotherapy (TTRNA-xALT) plus TTRNA-loaded dendritic cell vaccine.

Following surgical resection, biopsy, or cytology examination with confirmatory pathologic diagnosis, patients will be enrolled into Group A (high-dose chemotherapy or HDC) or Group B (non-myeloablative or NMA salvage chemotherapy) based on eligibility for HDC. Patients with localized relapse and have not failed HDC+ peripheral blood stem cell transplant (PBSCT) previously will be enrolled into Group A. Patients with disseminated disease, have previously failed HDC+PBSCT, or are otherwise considered poor candidates for HDC based on overall health status, but otherwise meet eligibility criteria, will be enrolled into Group B. All patients will receive DC + xALT therapy.

ELIGIBILITY:
Inclusion Criteria:

Screening:

* Age ≤ 30 years of age.
* Suspected first recurrence/progression of MB/PNET since completion of definitive focal +/- craniospinal irradiation. Disease progression prior to receiving definitive focal +/- craniospinal irradiation will not disqualify patients from enrollment if they have subsequently failed definitive radiotherapy and are at first recurrence/progression at time of enrollment. Patients who are unable to receive radiation therapy due to genetic disorders that put them at significant risk for radiation-induced secondary malignancies (i.e. Gorlin's syndrome or NF1 mutation) are eligible for enrollment at first disease recurrence/progression.

Re-MATCH Protocol:

* Patients must have histologically confirmed recurrent MB/PNET that is a first relapse/progression after completion of definitive radiotherapy +/- craniospinal irradiation. Patients with a first relapse/progression who are unable to receive radiation therapy due to genetic disorders that put them at significant risk for radiation-induced secondary malignancies (ie. Gorlin's syndrome or NF1 mutation) are eligible for enrollment.
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration.
* Karnofsky Performance Status of ≥ 50% or Lansky Performance Score of ≥ 50.
* Absolute Neutrophil Count (ANC) ≥ 1000/µl (unsupported).
* Platelets ≥ 100,000/µl (unsupported).
* Hemoglobin > 8 g/dL (may be supported).
* Serum creatinine ≤ upper limit of institutional normal
* Bilirubin ≤ 1.5 times upper limit of normal for age.
* Serum Glutamic Oxaloacetic Transaminase (ALT) ≤ 3 times institutional upper limit of normal for age.
* Serum Glutamic Oxaloacetic Transaminase (AST) ≤ 3 times institutional upper limit of normal for age.
* Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.
* Patient or patient guardian consent to peripheral blood stem cell (PBSC) and/or bone marrow harvest following registration if PBSC or bone marrow (CD34 count of at least 2x10^6/kg) has not been previously stored and available for use.
* Signed informed consent according to institutional guidelines must be obtained prior to registration.

Exclusion Criteria:

* Pregnant or need to breast feed during the study period.
* Active infection requiring treatment or an unexplained febrile (> 101.5F) illness.
* Known immunosuppressive disease, human immunodeficiency virus infection, or carriers of Hepatitis B or Hepatitis C virus.
* Patients with active renal, cardiac (congestive cardiac failure, myocardial infarction, myocarditis), or pulmonary disease.
* Patients receiving concomitant immunosuppressive agents for medical condition.
* Patients who need definitive radiotherapy for treatment of recurrent MB/PNET. Focal boost radiotherapy may be delivered prior to immunotherapy if required for local control.
* Patients receiving any other concurrent anticancer or investigational drug therapy.
* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction).
* Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2010-09-07 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2025-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duane Mitchell, MD, PhD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-six patients were assessed for eligibility in the Phase II trial. Ten subjects were excluded; seven did not meet eligibility and three declined participation prior to allocation to intervention arm.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 7 | 19
Completed | 7 | 15
Not Completed | 0 | 4
Not completed — progressed prior to vaccine | 0 | 2
Not completed — unable to make vaccine | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 7 | 15 | 22
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 15 [13.5 to 19] | 10 [6.5 to 14.5] | 12.5 [7.5 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 7 | 12 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 7 | 9 | 16
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 15 | 22

OUTCOME MEASURES:

1. Primary Outcome: 12 Month Progression-free Survival (PFS-12)
Description: PFS is defined as time interval from date of first DC vaccine to date of progression (death is also treated as progression) or censoring, whichever happens first.
Time Frame: up to 12 months
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 7 | 15
Days | 215 [110 to NA] — In Group A, we have insufficient participants with events. | 69 [41 to 151]
Statistical Analysis 1: Comparison: Group A; Based on published literature, PFS-12 for patients with recurrent disease after initiating treatment with HDC + PBSCT or standard salvage therapy was 33% (95% confidence interval of 10%, 59%). The study was designed to differentiate between a PFS-12 rate of 33% (null hypothesis) and 55% (alternative hypothesis). If 35 patients enrolled, this assessment has 90% power assuming a type I error rate of 0.10. We assume that PFS of historical controls follows exponential distribution; Test type: Superiority; p = 0.927, Log Rank — This is the p-value comparing Group A with historical control; One sample log rank; comparing two curves = 0.286, 90% CI 2-sided [0.107 to 0.764]
Statistical Analysis 2: Comparison: Group B; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Log Rank — This is the p-value comparing Group B with historical control; compare two curves = 0
Statistical Analysis 3: Comparison: Group A vs Group B; Test type: Superiority; p < 0.001, Log Rank — This is the p-value comparing Groups A and B combined with historical control; Comparing two curves = 0.091, 90% CI 2-sided [0.03 to 0.276]

2. Secondary Outcome: Objective Radiographic Response Rate
Description: Radiographic response will be assessed as a percentage change in tumor size from pre-treatment (baseline) MRI scans of the brain and spine obtained with and without contrast. Evaluation will be based on the NCI-endorsed, World Health Organization RECIST criteria and using a modified version of the MacDonald criteria (complete response, partial response, stable disease, progressive disease or not assessible).
Time Frame: best overall radiographic response through duration on study (up to 60 months)
Reporting Status: Not Posted

3. Secondary Outcome: Correlate Magnitude and Persistence of Anti-tumor Humoral or Cellular Immunity With Clinical Outcome
Description: Peripheral blood will be used to compare pre-therapy lymphocyte function to defined intervals after each immunization. Blood will be obtained for immunologic monitoring prior to non-mobilized leukapheresis, prior to immunotherapy, 1 day post Vaccine #1, 4 (+/- 1) days post Vaccine #1, weekly post Vaccine #1 for six weeks.
Time Frame: baseline compared to 6 weeks post vaccine #1 and longitudinal measures through overall survival (up to 60 months)
Reporting Status: Not Posted

4. Secondary Outcome: Evaluate Changes in Cytokine Profile and Toll-Like Receptor Activation Status
Description: We will measure serum cytokines pre and post therapy. Blood will be obtained for immunologic monitoring prior to non-mobilized leukapheresis, prior to immunotherapy, 1 day post Vaccine #1, 4 (+/- 1) days post Vaccine #1, weekly post Vaccine #1 for six weeks.
Time Frame: baseline compared to 6 weeks post vaccine #1 and longitudinal measures through overall survival (up to 60 months)
Reporting Status: Not Posted

5. Secondary Outcome: Characterize Immunologic Phenotype of Lymphocyte Subsets and NK Cells
Description: We will conduct flow cytometry from patient samples. Blood will be obtained for immunologic monitoring prior to non-mobilized leukapheresis, prior to immunotherapy, 1 day post Vaccine #1, 4 (+/- 1) days post Vaccine #1, weekly post Vaccine #1 for six weeks.
Time Frame: baseline compared to 6 weeks post vaccine #1 and longitudinal measures through overall survival (up to 60 months)
Reporting Status: Not Posted

6. Secondary Outcome: Determine of Overall Survival Rate
Description: Kaplan-Meier estimator will be used to describe length of overall survival from initiation of vaccine #1 for both Groups A and B.
Time Frame: up to 60 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: There are two AE periods. The first begins at initiation of non-mobilized leukapheresis and ends 24 hrs after completion of the procedure. The second starts with initiation of consolidation or NMA chemotherapy and continues until 100 days after either the infusion of PBSCs or completion of chemotherapy for subjects not receiving PBSCs. AEs are not collected from the end of the leukapheresis period until the start of consolidation/NMA chemotherapy when subjects received salvage chemotherapy.
Description: An "AE" will be defined as any adverse change from the subject's pre-treatment baseline condition, including any clinical or laboratory test abnormality that occurs during the course of research after treatment has started. A summary of recorded AEs will be kept which will categorize the event by organ system, relationship to treatment, its grade of severity, and resolution.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 6/7 | 17/19
Serious Adverse Events (participants affected / at risk) | 4/7 | 5/19
Other Adverse Events (participants affected / at risk) | 7/7 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=7) | Group B (N=19)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Colitis, Infectious (Infections and infestations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Metabolic Acidosis
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=7) | Group B (N=19)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Increased ALT (Investigations) | 1 (4) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 7 (19) | 10 (25)
Anorexia (Metabolism and nutrition disorders) | 5 (7) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (3) | 2 (2)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2)
Blurred vision (Eye disorders) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 2 (3) | 0 (0)
Confusion (Nervous system disorders) | 2 (2) | 0 (0)
Decreased platelet count (Blood and lymphatic system disorders) | 4 (5) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (2)
Enterocolitis (Infections and infestations) | 1 (1) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Fever (General disorders) | 4 (6) | 2 (4)
Headache (Nervous system disorders) | 1 (2) | 1 (1)
hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
hypomagnesemia (Metabolism and nutrition disorders) | 1 (3) | 1 (3)
hypophosphatemia (Metabolism and nutrition disorders) | 4 (5) | 1 (5)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 5 (12) | 9 (23)
Lymphocyte count decreased (Investigations) | 6 (16) | 14 (28)
Mucositis oral (Gastrointestinal disorders) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8) | 4 (6)
neutrophil count decreased (Investigations) | 5 (13) | 12 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 3 (22) | 5 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain - access site (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (5) | 3 (5)

LIMITATIONS AND CAVEATS:
Given that number evaluable subjects was below targeted enrollment, this study was underpowered for the desired statistical comparison.

Due to COVID we anticipate that the immunologic secondary endpoints will be completed in 6-12 months or change to exploratory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT01326104/Prot_SAP_000.pdf